CLINICAL TRIAL: NCT04005599
Title: Magnesium Sulfate in Substitution to Remifentanil. Intra-operative Analgesia Assessed by the Surgical Stress Index. Randomized and Blind Clinical Trial
Brief Title: Opioid Sparing General Venous Anesthesia With Magnesium Sulfate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Joaquim Edson Vieira, Associate professor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAAE 12614719.1.0000.0068
Record Dates: First submitted 2019-06-25; First posted 2019-07-02 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Magnesium Sulfate; Postoperative Pain; Opioid Use
Keywords: Postoperative pain; opioid; Postoperative analgesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Prospective, controlled, randomized and double-blind clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The anesthesiologist in charge of randomization will number 40 opaque envelopes and insert a card in each with the corresponding information of the group (according to the lottery) and the medication to be administered. Another anesthesiologist in charge of preparing the blind solution alone will open the envelope. Both of these investigators, as well as the anesthesiologist providing anesthesia and the anesthesiologist in charge of data evaluation will not participate in any of the other steps of the trial. The patients will be blinded to their own treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remifentanil group (Active Comparator): Intravenous anesthesia with propofol and remifentanil
  Interventions: Drug: Remifentanil group
- Magnesium group (Experimental): Intravenous anesthesia with propofol and magnesium sulfate
  Interventions: Drug: Magnesium sulfate group

INTERVENTIONS:
Drug: Remifentanil group — Venous general anesthesia with propofol and remifentanil.
  Arms: Remifentanil group
Drug: Magnesium sulfate group — Venous general anesthesia with propofol and magnesium sulfate
  Arms: Magnesium group

SUMMARY:
Magnesium sulfate has been shown to be useful in many situations in medicine, such as eclampsia prevention and treatment, pulmonary hypertension, arterial pressure, asthma, cardiac arrhythmias and pheochromocytoma. Recently there has been a growing a big interest in this drug as an useful adjuvant in anesthesia, with analgesic and anesthetic sparing effect, antihyperalgesic property and potentialization of the neuromuscular blocker agent effect. On the other hand there has been a growing concern related to opioid administration, such as hyperalgesia, delayed return of intestinal function and the (still controversial) possibility of facilitating effect on tumor growth and metastases in cancer patients.

This project is based on a previous randomized, double blind prospective trial (conducted by one of these authors and not yet published) comparing two groups of patients who received general intravenous total anesthesia with propofol in controlled target infusion.

The surgical stress index is obtained by the interaction between the interval between heart beats and the amplitude of the photoplethysmography wave, whose algorithm generates a number related to the hemodynamic result of the increase of the sympathetic tone, which has shown to be the most sensitive resource in detecting the imbalance between the stimulus nociceptive and anti-nociception.

DETAILED DESCRIPTION:
Magnesium sulfate has been shown to be useful in many situations in medicine, such as eclampsia prevention and treatment, pulmonary hypertension, arterial pressure, asthma, cardiac arrhythmias and pheochromocytoma. Recently there has been a growing a big interest in this drug as an useful adjuvant in anesthesia, with analgesic and anesthetic sparing effect, antihyperalgesic property and potentialization of the neuromuscular blocker agent effect. On the other hand there has been a growing concern related to opioid administration, such as hyperalgesia, delayed return of intestinal function and the (still controversial) possibility of facilitating effect on tumor growth and metastases in cancer patients.

This project is based on a previous randomized, double blind prospective trial (conducted by one of these authors and not yet published) comparing two groups of patients who received general intravenous total anesthesia with propofol in controlled target infusion.

The surgical stress index is obtained by the interaction between the interval between heart beats and the amplitude of the photoplethysmography wave, whose algorithm generates a number related to the hemodynamic result of the increase of the sympathetic tone, which has shown to be the most sensitive resource in detecting the imbalance between the stimulus nociceptive and anti-nociception.

Objectives The main objective of this project is to evaluate the feasibility of the use of magnesium sulfate in replacement of remifentanil as the main analgesic agent in total venous general anesthesia in patients submitted to post-bariatric dermolipectomy surgery.

The secondary objectives will be comparison of propofol consumption, time to onset of action, time of action and cisatracurium consumption between groups. We will evaluate pain scores in the immediate postoperative period and in the mornings and afternoons of the 3 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 60 year-old
* body mass index < 35 kg/m²
* American Society of Anesthesiologists score < III
* agreement to participate and sign the informed consent form.

Exclusion Criteria:

* Allergy to any medications of the trial
* neuromuscular diagnosed disorder
* cardiac conduction blockade (atrioventricular block II or higher),
* use of illicit drugs
* use of calcium channel blockers
* creatinine > 2 mg/dl.

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2022-01-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of using magnesium sulfate as analgesic of venous general anesthesia | Surgery time
  Changes in systolic blood pressure (mmHg) after tracheal intubation and surgical incision in both groups.

SECONDARY OUTCOMES:
Anesthetic consumption. | During surgery
  Consumption of propofol (mg) and cisatracurium.
Neuromuscular blocker action | During surgery
  Onset and offset of cisatracurium (minutes)
Postoperative pain | Three days
  Pain scores (verbal numerical scale from 0 to 10).

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim Vieira, Professor, Principal Investigator — University of Sao Paulo School of Medicine
Locations (1):
- Hospital das Clínicas - Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
We have no plan to made individual participant data available to other researchers.